CLINICAL TRIAL: NCT06252038
Title: Rural Alliance for Diabetes Prevention
Acronym: RAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Kansas State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00150103; R01DK132362 (NIH)
Record Dates: First submitted 2024-01-12; First posted 2024-02-09 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: PreDiabetes
Keywords: Diabetes Prevention Program; HbA1c; Physical Activity; Weight Loss
MeSH Terms: conditions — Prediabetic State; Motor Activity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Video Diabetes Prevention Program (Experimental): Participants randomized to the group video DPP for 12-months.
  Interventions: Behavioral: Zoom Group Video (GV)
- Self Directed Diabetes Prevention Program (Active Comparator): Participants randomized to the self directed DPP for 12-months.
  Interventions: Behavioral: Self Directed (SD)

INTERVENTIONS:
Behavioral: Zoom Group Video (GV) — Zoom delivery of the DPP. Participants have access to Prevent T2 Curriculum and connected technology to track weight and physical activity.
  Arms: Group Video Diabetes Prevention Program
Behavioral: Self Directed (SD) — Self directed delivery of the DPP. Participants have access to online curriculum, lifestyle coach and connected technology to track weight and physical activity.
  Arms: Self Directed Diabetes Prevention Program

SUMMARY:
The purpose of this randomized controlled trial is to compare the effectiveness of Cooperative Extension implementing two delivery methods (group video vs. self-directed) and participant recruitment strategies of the National Diabetes Prevention Program (NDPP) to adults in rural communities. Exploratory assessments of implementation facilitators and barriers will be completed to determine strategies that may impact intervention effectiveness and that may support or impede the implementation, dissemination, and effectiveness of Cooperative Extension to deliver the NDPP to prediabetic adults in rural areas.

DETAILED DESCRIPTION:
This 12 mo. Type II hybrid effectiveness-implementation trial will compare effectiveness (weight loss, physical activity, HbA1c) of Cooperative Extension delivering the Diabetes Prevention Program (DPP) by group video using Zoom® (GV) vs. a self-directed (SD) control. Active vs. passive participant recruitment strategies will be compared on recruitment outcomes including time to full enrollment, participant yield, and retention rates. Ten Cooperative Extension local units/districts serving rural Kansas counties will be allocated to either active or passive recruitment. Each of the sites will recruit adults with prediabetes living in the county served by Kansas State Research and Extension site and will be randomized to one of the 2 intervention arms. A centralized team of Cooperative Extension Agents who complete NDPP lifestyle coach training will serve as interventionists for both the GV and SD arms. Primary (weight) and secondary outcomes (HbA1c, the proportion of participants meeting weight loss (≥ 5%) and physical activity goals (≥150 min./wk.) will be assessed at baseline, 6 and 12 mos. Findings will inform best practices in the delivery of the DPP through Cooperative Extension in rural communities that could reach this high risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* BMI ≥25 kg/m2, ≥23 kg/m2 if Asian
* Blood test results in the pre diabetic range within the last year (HbA1C = 5.7%-6.4% or fasting plasma glucose= 100-125 mg/dl or 2-hr. plasma glucose following a 75-gm glucose load = 140-199 mg/dL) or have previous diagnosis of gestational diabetes or a positive screening for pre diabetes based on CDC pre diabetes risk test
* Willing to travel to KSRE site for orientation and outcome testing
* Available to attend pre-specified meeting time of GV for their respective KSRE location
* Medically stable as deemed by primary care provider consent
* English speaking

Exclusion Criteria:

* Previous diagnosis of Type I or II diabetes
* Taking FDA-approved weight loss medications
* Primary care provider stating that patient should not participate
* Self-report as currently pregnant or within 6 weeks of having given birth (or planning to become pregnant in the next 12 months)
* Unable to engage in physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Weight change across 12 months | Baseline to 12 months
  Weight (kg) will be assessed to the nearest 0.1 kg with a calibrated scale (Belfour Inc., Model #PS6600). All participants will be weighed between the hours of 6 and 10 am following an overnight fast of at least 8 hours in a standard hospital gown.

SECONDARY OUTCOMES:
HbA1c change across 12 months | Baseline to 12 months
  Hemoglobin A1c will be collected and assessed by Quest Diagnostic. Participants will be required to fast for at least 12 hours before blood draw. A total of 3-5 teaspoons of blood will be collected by inserting a needle in a vein in the arm for routine laboratory tests at each clinic visit. Participant blood samples will be used to measure HbA1c.
CDC-NDPP Weight Loss Goal | Baseline to 12 months
  CDC-NDPP weight loss goal will be categorized as the percentage of participants who achieve ≥ 5% weight loss across the 12 month intervention.
CDC-NDPP Physical Activity Goal | Baseline to 12 months
  CDC-NDPP physical activity goal will be categorized by the percentage of participants who achieve an average of ≥ 150 min./wk. of PA across the 12 month intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Gorczyca, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No